CLINICAL TRIAL: NCT07328334
Title: Longitudinal Assessment of Maximal Inspiratory Pressure and Functional Capacity Following Inspiratory Muscle Training in Frail Older Adults: A Randomized, Double-Blind, Sham-Controlled Trial
Brief Title: Longitudinal Assessment of Maximal Inspiratory Pressure and Functional Capacity Following Inspiratory Muscle Training in Frail Older Adults (IMT-2)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Francisco de Vitoria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UFV-IMT2
Record Dates: First submitted 2025-12-19; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Frailty Syndrome; Geriatric Health; Respiratory Muscle Weakness; Age-Related Frailty
Keywords: Inspiratory Muscle Training; Diaphragm Ultrasound; Older Adults
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory Muscle Training (Experimental): Participants perform an 8-week inspiratory muscle training program using a threshold device (PowerBreathe). Training consists of 30 inspirations, once daily, 5 days per week. The initial load is set at 50% of each participant's maximal inspiratory pressure (MIP) and is increased weekly by 5 cmH#O up to 80% of MIP. All sessions are supervised by healthcare professionals, with continuous monitoring of oxygen saturation and heart rate
  Interventions: Device: Inspiratory Muscle Training
- Inspiratory Muscle Training (Sham) (Sham Comparator): Participants follow the same 8-week training schedule using the threshold device (PowerBreathe), but with a constant load of 15% of maximal inspiratory pressure (MIP) and no weekly progression. Training consists of 30 inspirations, once daily, 5 days per week. The procedure mimics the experimental intervention but provides minimal physiological stimulus. All sessions are supervised, with monitoring of oxygen saturation and heart rate
  Interventions: Device: Sham Inspiratory Muscle Training

INTERVENTIONS:
Device: Inspiratory Muscle Training — Participants perform 30 breaths once daily, 5 days per week for 8 weeks using a threshold inspiratory muscle training device. The load begins at 50% of maximal inspiratory pressure (MIP) and increases by 5 cmH#O weekly up to 80% of MIP. Sessions are supervised and oxygen saturation and heart rate are monitored.
  Arms: Inspiratory Muscle Training
Device: Sham Inspiratory Muscle Training — Participants use the same device and schedule as the experimental group (30 breaths once daily, 5 days per week for 8 weeks) but with a constant load of 15% of maximal inspiratory pressure (MIP), with no weekly progression. This mimics the procedure while providing minimal physiological stimulus. Supervision and monitoring are identical to the experimental arm.
  Arms: Inspiratory Muscle Training (Sham)

SUMMARY:
This study aims to evaluate the effects of an 8-week inspiratory muscle training program on maximal inspiratory pressure and functional capacity in frail older adults aged 80 years and above. Frailty is associated with reduced physical capacity, declines in functional performance, impaired respiratory performance, and a higher risk of disability. Inspiratory muscle training is a simple, low-cost intervention that may improve breathing function, inspiratory muscle strength, and overall health in very old adults, but evidence in this age group remains limited.

Participants will be randomly assigned to one of two groups: a high-load inspiratory muscle training group or a low-load sham training group. Both groups will use a threshold device and perform 30 breaths once per day, five days per week, for eight weeks. The experimental group will train with progressively increasing resistance (50% to 80% of maximal inspiratory pressure), while the sham group will use a minimal and non-progressive load (15% of maximal inspiratory pressure). All sessions will be supervised and monitored for safety.

The main goal of the study is to determine whether inspiratory muscle training improves maximal inspiratory pressure (MIP), an established measure of global inspiratory muscle strength. Secondary outcomes include measures of functional capacity, reflecting the ability to perform physical tasks relevant to daily living in very old adults. These outcomes will allow the evaluation of the clinical relevance of improvements in inspiratory muscle strength in this population.

Assessments will be performed before the intervention, immediately after the 8-week program, and again at one and three months after the end of the intervention to examine both immediate and short-term effects. This study may contribute valuable evidence regarding the safety, feasibility, and clinical benefits of inspiratory muscle training in frail very old adults, particularly its impact on inspiratory muscle strength and functional capacity, supporting its potential implementation in rehabilitation and geriatric care.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 80 years or older.
* Clinical diagnosis of frailty, defined by a Short Physical Performance Battery (SPPB) score < 9.
* Ability to stand and walk with or without assistive devices.
* Ability to understand and follow instructions for inspiratory muscle training.
* Stable medical condition for at least 3 months prior to enrollment.
* Capacity to provide informed consent or availability of a legal

Exclusion Criteria:

* Acute or unstable cardiovascular, respiratory, or metabolic conditions.
* Severe cognitive impairment that prevents understanding the procedures.
* Diagnosis of neuromuscular diseases affecting respiratory muscles (e.g., ALS, myopathies).
* Severe or uncontrolled hypertension (≥180/110 mmHg).
* Recent thoracic or abdominal surgery (<3 months).
* Severe musculoskeletal disorders limiting participation in training.
* History of recurrent syncope, severe dizziness, or intolerance to respiratory maneuvers.
* Any condition judged by the research team to compromise safety or participation.

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09-10 (Estimated)

PRIMARY OUTCOMES:
Maximal Inspiratory Pressure (MIP) | Before-intervention; Immediately after intervention; 1-month after intervention; 3 months after intervention
  Maximal Inspiratory Pressure (MIP) will be measured using a calibrated handheld manometer following standardized respiratory assessment guidelines. Participants will be instructed to perform a maximal inspiratory effort from residual volume through the mouthpiece with their nose occluded. At least three maneuvers will be recorded, ensuring less than 10% variability between attempts. The highest reproducible value (cmH₂O) will be used for analysis. This measure reflects global inspiratory muscle strength and is widely validated in older and frail populations.
Six-Minute Walk Test (6MWT) | Before-intervention; Immediately after intervention; 1-month after intervention; 3 months after intervention
  Functional exercise capacity will be assessed using the Six-Minute Walk Test (6MWT). Participants will be instructed to walk at their fastest possible pace for six minutes along a 30-meter corridor, covering the greatest distance possible. The total distance walked (in meters) will be recorded.
  Participants will be continuously accompanied by the therapist and may use assistive devices and/or supplemental oxygen if required.
Timed Up and Go Test (TUG) | Before-intervention; Immediately after intervention; 1-month after intervention; 3 months after intervention
  Functional mobility and fall risk will be evaluated using the Timed Up and Go (TUG) test. Participants will start seated in a chair with armrests. On command, they will stand up, walk 3 meters, turn around, return to the chair, and sit down. The total time to complete the task will be recorded in seconds.
  Interpretation criteria:
  < 20 seconds: normal performance
  ≥ 20 seconds: increased risk of falls
Five Times Sit-to-Stand Test (5STS) | Before-intervention; Immediately after intervention; 1-month after intervention; 3 months after intervention
  Lower limb functional strength will be assessed using the Five Times Sit-to-Stand Test (5STS). Participants will sit on a 43-45 cm high chair without armrests, with arms crossed over the chest, and will be instructed to stand up and sit down five times as quickly as possible.
  The total time to complete the test will be recorded in seconds. The minimal detectable change ranges from 3.6 to 4.2 seconds, and the minimal clinically important difference is 2.3 seconds. Age-related normative values will be considered for interpretation.
Upper Limb Muscle Strength (Handgrip Dynamometry) | Before-intervention; Immediately after intervention; 1-month after intervention; 3 months after intervention
  Upper limb muscle strength will be assessed using handgrip dynamometry following the recommendations of the American Society of Hand Therapists. Participants will be seated with the shoulder in adduction and neutral rotation, the elbow flexed at 90°, the forearm in neutral position, and the wrist positioned between 0° and 30° of extension.
  Three maximal grip strength measurements will be obtained from the dominant hand, with 1 minute of rest between trials. The highest value will be selected for analysis. Handgrip strength will be measured using a JAMAR dynamometer (Lafayette Instrument, Lafayette, IN, USA).
Lower Limb Muscle Strength (Isometric Knee Extension Dynamometry) | Before-intervention; Immediately after intervention; 1-month after intervention; 3 months after intervention
  Lower limb muscle strength will be assessed using isometric dynamometry to evaluate maximal voluntary contraction (MVC) of the knee extensors. The protocol described by Hung et al. will be followed. Participants will perform two maximal isometric contractions, each lasting 5 seconds, with 3 minutes of rest between contractions to allow phosphocreatine resynthesis.
  Participants will be seated at the edge of a physiotherapy table with the knee positioned at 90° of flexion. The dynamometer will be placed at the level of the malleoli to standardize the lever arm and ensure maximal isometric contraction. The peak force achieved during each contraction will be recorded and normalized to body weight, with results expressed in Newtons (N).
  Lower limb dynamometry will be performed using the ActiveForce 2 device (Activbody, San Diego, CA, USA).
Muscle Oxygenation | Before-intervention; Immediately after intervention; 1-month after intervention; 3 months after intervention
  Muscle oxygen saturation (SmO₂) will be assessed using the Moxy Monitor (Fortiori Design LLC, Hutchinson, MN, USA), a wireless and portable device based on near-infrared spectroscopy (NIRS).
  The measurement protocol described by Contreras-Briceño et al. will be followed and will consist of a 180-second resting measurement, followed by continuous monitoring during the Six-Minute Walk Test (6MWT).
  Outcome values will correspond to the mean SmO₂ (%) recorded during the final 30 seconds of each phase.
  The sensor will be placed over the muscle belly of the vastus lateralis following standard NIRS placement recommendations.
Total Hemoglobin Concentration (THb) | Before-intervention; Immediately after intervention; 1-month after intervention; 3 months after intervention
  Total hemoglobin concentration (THb) will be assessed using the same NIRS device (Moxy Monitor, Fortiori Design LLC, Hutchinson, MN, USA).
  Data acquisition and analysis will be performed using dedicated software (Moxy Software v1.5.5; Idiag, Fehraltorf, Switzerland). The same protocol will be applied: a 180-second resting measurement followed by continuous monitoring during the Six-Minute Walk Test (6MWT).
  Outcome values will correspond to the mean THb values recorded during the final 30 seconds of each phase.
  The sensor placement will be identical to that used for SmO₂ assessment (vastus lateralis).

IPD SHARING:
Plan to Share IPD: Undecided
At this time, it is unclear whether individual participant data (IPD) will be shared.
  Data sharing will depend on institutional policies, ethical approvals, participant privacy considerations, and the feasibility of preparing de-identified datasets. A final decision will be made once data collection and analysis are completed.